CLINICAL TRIAL: NCT01618955
Title: Phase 2, Multi-Center, Open-Label, Single-Dose, Single Arm, In-Clinic Study to Evaluate the Actual Human Use of Methotrexate Subcutaneously Administered Via the VIBEX™ MTX Auto-Injector Device in Adult Patients With Rheumatoid Arthritis.
Brief Title: Actual Human Use of Methotrexate (MTX) Subcutaneously Administered Via the VIBEX™ MTX Auto-Injector Device
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTX-11-002
Record Dates: First submitted 2012-06-04; First posted 2012-06-14 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VIBEX MTX (Active Comparator): VIBEX MTX dose based on the subject's current therapeutic regimen of MTX and rheumatoid arthritis disease status
  Interventions: Device: VIBEX MTX

INTERVENTIONS:
Device: VIBEX MTX — Self-administration of Single Dose of SC MTX using Vibex MTX 10 mg, 15 mg, 20 mg or 25 mg Device
  Other Names: prefilled autoinjector device

SUMMARY:
The purpose of this study is to assess the usability of the VIBEX MTX device for SC self-injection of methotrexate.

DETAILED DESCRIPTION:
Primary objective:

- To assess the safe usability of the VIBEX MTX device for subcutaneous (SC) self-injection of methotrexate (MTX) in adult patients with rheumatoid arthritis (RA) after standardized training by site personnel and review of written instructions

Secondary objectives:

* To evaluate the reliability and robustness of the VIBEX MTX device
* To evaluate the safety and local tolerance of an SC self-injection of MTX using the VIBEX MTX device
* To evaluate the effectiveness and ease of use of the VIBEX MTX device patient education tools for SC self-injection

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age, diagnosed with Rheumatoid Arthritis

Exclusion Criteria:

* Pregnant females
* Any other clinically significant disease or disorder which, in the opinion of the investigator might put the subject at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Kivitz, MD;CPI, Principal Investigator — Altoona Center for Clinical Research
Locations (1):
- Altoona Center for Clinical Research, Duncansville, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened & enrolled at 8 sites in the US. There were 20 subjects in 10mg, 30 subjects in 15mg, 31 subjects in 20mg and 20 subjects in 25mg dose group. The dose group was determined by the Investigator based on subject's current therapeutic regimen of MTX and disease status. The patient's dose was the same for the entire study.
Pre-assignment Details: All patients received standardized subcutaneous self-injection training per Instructions For Use, then demonstrated the self-injection procedure with practice device and completed the training confirmation questionnaire. And then the subjects were allowed to self-administer the study dose via Vibex MTX.
Groups:
- MTX 10 mg; MTX 15 mg; MTX 20 mg; MTX 25 mg: Self-administration of Subcutaneous Methotrexate using VIBEX MTX
Period: Overall Study
Arm/Group | MTX 10 mg | MTX 15 mg | MTX 20 mg | MTX 25 mg
Started | 20 | 30 | 31 | 20
Completed | 20 | 30 | 31 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 101 patients were included in the Safety Population, which consisted of all patients who received study drug and administered a successful or unsuccessful self-injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | MTX 10 mg | MTX 15 mg | MTX 20 mg | MTX 25 mg | Total
Number analyzed (Participants) | 20 | 30 | 31 | 20 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (11.46) | 61.8 (9.00) | 59.5 (10.46) | 59.1 (9.92) | 60.9 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 26 | 16 | 80
  Male | 2 | 10 | 5 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 1 | 7
  White | 18 | 29 | 27 | 19 | 93
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 19 | 29 | 30 | 20 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 30 | 31 | 20 | 101
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.4 (7.54) | 31.3 (7.26) | 30.5 (6.46) | 30.3 (5.28) | 30.9 (6.64)

OUTCOME MEASURES:

1. Primary Outcome: Safe Usability of the VIBEX MTX Device for Subcutaneous (SC) Self-injection With Methotrexate (MTX) in Adult Patients With Rheumatoid Arthritis (RA) as Demonstrated by Successful Self-Injection
Description: A total of 101 patients were included in the Safety Population, which consisted of all patients who received standardized training by site personnel and review of written instructions. And then self-administered study drug using Vibex MTX device.
  The Assessment of Essential Tasks Questionnaire was completed by site personnel documenting a patient's performance of essential self-injection steps, including the following:
  1. SC self-injection was administered by the patient
  2. SC self-injection was intentional
  3. self-injection was administered in an appropriate location on the abdomen
  4. patient removed cap marked "1"
  5. patient removed cap marked "2"
  6. patient held device at injection site for 3 seconds
  7. patient confirmed that the window was obstructed
Time Frame: 24 hours
Population: The safety population consisted of all subjects who received study drug and administered a successful or unsuccessful self-injection. For categorical data, percentages are presented.
Measure: Number; unit: Percentage of Participants
Groups:
- Vibex MTX 10 mg; Vibex MTX 15 mg; Vibex MTX 20 mg; Vibex MTX 25 mg: Self-administration of subcutaneous methotrexate using Vibex MTX
Arm/Group | Vibex MTX 10 mg | Vibex MTX 15 mg | Vibex MTX 20 mg | Vibex MTX 25 mg
Number analyzed (Participants) | 20 | 30 | 31 | 20
Percentage of Participants
  SC self-injection was administered by patient (%) | 100 | 100 | 100 | 100
  SC self-injection was intentional (%) | 100 | 100 | 100 | 100
  SC self-injection was in abdomen (%) | 100 | 100 | 100 | 100
  Patient removed cap marked "1" (%) | 100 | 100 | 100 | 100
  Patient removed cap marked "2" (%) | 100 | 100 | 100 | 100
  Patient held device at injection site > 3 sec (%) | 100 | 100 | 100 | 100
  Patient confirmed that window was obstructed (%) | 100 | 100 | 100 | 100

2. Secondary Outcome: Reliability and Robustness of Vibex MTX Device as Well as Effectiveness of Patient Education Tools
Description: A total of 101 patients were included in the Safety Population, which consisted of all patients who received standardized training by site personnel and review of written instructions. And then self-administered study drug using Vibex MTX device
  1. Ease of use Questionnaire was completed by patients immediately after self-injection
  2. Training confirmation questionnaire was completed by patients after the training and then reviewed with PI or site coordinator
Time Frame: 24 hours
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Vibex MTX 10 mg | Vibex MTX 15 mg | Vibex MTX 20 mg | Vibex MTX 25 mg
Number analyzed (Participants) | 20 | 30 | 31 | 20
Percentage of Participants
  Device was easy to use (%) | 95 | 100 | 97 | 100
  Understood the written instructions (%) | 100 | 100 | 100 | 100
  Written instructions were clear & easy to follow % | 100 | 100 | 100 | 100
  Understood the training provided by site staff (%) | 100 | 100 | 100 | 100
  Training by site staff-clear & easy to follow (%) | 100 | 100 | 100 | 100
  Training Confirmation Questions answered right (%) | 90 | 93.3 | 96.8 | 95.0

3. Secondary Outcome: Safety of Vibex MTX Device
Description: A total of 101 patients were included in the Safety Population, which consisted of all patients who received standardized training by site personnel and review of written instructions. And then self-administered study drug using Vibex MTX device
  Injection site assessments were done 0.25 hour, 1 hour, 6 hours and 24 hours after an injection and reported as the following:
  * Erythema - 0 = None
  * Erythema - 1 = Very slight, barely perceptible
  * Erythema - 2 = Obvious, but well defined
  * Erythema - 3 = Moderate to severe
  * Erythema - 4 = Severe
Time Frame: 24 hours
Population: The safety population consisted of all subjects who received study drug and administered a successful or unsuccessful self-injection. For categorical data, counts and percentages are presented.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vibex MTX 10 mg | Vibex MTX 15 mg | Vibex MTX 20 mg | Vibex MTX 25 mg
Number analyzed (Participants) | 20 | 20 | 31 | 20
Percentage of Participants
  No Erythema at all post-dose time points (%) | 95 | 88.3 | 96.0 | 90.0
  Erythema very slight - barely perceptible (%) | 5 | 11.7 | 4.0 | 10.0

4. Secondary Outcome: Tolerance of Vibex MTX Device (Injection Site Pain Severity as Reported by Patient on VAS Scale - 0 mm = no Pain to 100 mm = Very Severe Pain)
Description: A total of 101 patients were included in the Safety Population, which consisted of all patients who received standardized training by site personnel and review of written instructions. And then self-administered study drug using Vibex MTX device.
  Visual Analog Scale assessment of injection site pain was reported by patients on 100 mm line immediately after an injection and at 24 hours after injection.
Time Frame: 24 hours
Population: The safety population consisted of all subjects who received study drug and administered a successful or unsuccessful self-injection. For continuous data, summary statistics (N, mean, standard deviation, median, minimum, and maximum) were provided.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Vibex MTX 10 mg | Vibex MTX 15 mg | Vibex MTX 20 mg | Vibex MTX 25 mg
Number analyzed (Participants) | 20 | 30 | 31 | 20
mm
  Severity of pain immediately after self-injection | 1.0 (1.05) | 7.6 (15.60) | 2.2 (2.91) | 2.4 (2.56)
  Severity of pain at 24 hours after self-injection | 1.7 (4.48) | 2.0 (4.15) | 1.0 (1.60) | 1.0 (1.23)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Vibex MTX 10 mg | Vibex MTX 15 mg | Vibex MTX 20 mg | Vibex MTX 25 mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/30 | 0/31 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/30 | 1/31 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibex MTX 10 mg (N=20) | Vibex MTX 15 mg (N=30) | Vibex MTX 20 mg (N=31) | Vibex MTX 25 mg (N=20)
Sick Sinus Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibex MTX 10 mg (N=20) | Vibex MTX 15 mg (N=30) | Vibex MTX 20 mg (N=31) | Vibex MTX 25 mg (N=20)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less